CLINICAL TRIAL: NCT07208097
Title: Stereotactic Thrombolysis With Tenecteplase for Supratentorial Intracerebral Hemorrhage
Acronym: STEPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Tang Zhouping, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB202511008
Record Dates: First submitted 2025-04-08; First posted 2025-10-06 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-09

CONDITIONS: Intracerebral Haemorrhage; Minimally Invasive Treatment
Keywords: intracerebral haemorrhage; minimally invasive treatment; hematoma evacuation; tenecteplase
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Tenecteplase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MIS+TNK (Experimental): In this group, patients receive standard medical treatment plus stereotactic minimally invasive aspiration combined with tenecteplase. The single dose of tenecteplase is 0.5mg.
  Interventions: Procedure: Stereotactic thrombolysis with Tenecteplase
- Standard medical treatment (No Intervention): Patients randomized to the control group will receive standard medical management according to the 2022 AHA/ASA Guideline for the Management of Spontaneous Intracerebral Hemorrhage.

INTERVENTIONS:
Procedure: Stereotactic thrombolysis with Tenecteplase — Stereotactic thrombolysis with Tenecteplase for ICH is a minimally invasive method for evacuation hematoma. The hematoma puncture target is identified via CT imaging before surgery. After local anesthesia and sedation, stereotactic minimally invasive surgery is performed with the Leksell stereotactic frame. A postoperative CT scan is immediately conducted to confirm the absence of intracranial rebleeding before administering tenecteplase into the hematoma. Tenecteplase is fully diluted in 2 mL of saline and injected into the hematoma cavity via an irrigation catheter. The drainage tube is clamped for 1 hour before opening (early opening is permitted if necessary). The single dose of TNK is 0.5 mg and can be administered with a maximum of 2 dose in every 24 hours. The target hematoma clearance criteria is: residual hematoma volume ≤10 mL or ≤20% of the initial volume.
  Arms: MIS+TNK

SUMMARY:
This is an phase III prospective, multi-center, open-label, randomized controlled trial (RCT) with blinded endpoint assessment. It plans to enroll 768 subjects with spontaneous supratentorial intracerebral hemorrhage, who will be randomly assigned in a 1:1 ratio to the investigational arm (stereotactic minimally invasive puncture for intracerebral hemorrhage combined with TNK liquefaction drainage, single TNK dose of 0.5mg per time or the standard medical treatment group.

DETAILED DESCRIPTION:
Intracerebral hemorrhage (ICH) is an acute cerebrovascular disease with an incidence rate of 60-80 cases per 100,000 population annually, accounting for approximately 10%-20% of all strokes. Early mortality in ICH patients can reach 30%-40%, and the disability rate remains high in later stages, with roughly two-thirds of patients ultimately dying or becoming disabled.

Brain injury caused by ICH can be categorized into primary and secondary damage. Primary injury results from direct trauma to white matter tracts, the blood-brain barrier, and hematoma mass effect immediately following bleeding. Secondary injury arises from mechanisms such as inflammation, blood-brain barrier disruption, cerebral edema, perihematomal edema, cytotoxicity, and oxidative stress, leading to neurological deficits. Clinical studies have confirmed that hematoma removal reduces mortality in ICH patients and may improve neurological outcomes. Minimally invasive hematoma evacuation combined with thrombolytics like rt-PA or urokinase has shown safety and reduced mortality but fails to improve functional outcomes. Post-hoc analyses reveal variable efficacy of rt-PA in liquefying hematomas, with incomplete evacuation and residual clots in some patients. Theoretically, faster and more efficient hematoma liquefaction could enhance clinical outcomes. Tenecteplase has demonstrated superior efficacy, rapid action, and safety in ischemic stroke compared to rt-PA, suggesting potential benefits for ICH hematoma clearance.

To determine the efficacy and safety of local injection of TNK via stereotactic minimally invasive puncture surgery for the treatment of acute spontaneous supratentorial intracerebral hemorrhage (ICH). This is a national, multicenter clinical trial spontaneously organized and designed by the investigators. It employs a Phase III prospective, multicenter, open-label, randomized, standard medical therapy parallel-controlled design, with blinded endpoint assessors. Subjects meeting the inclusion and exclusion criteria will be enrolled according to randomization principles. Investigators blinded to group allocation will conduct assessments and evaluations at various time points during the follow-up period for enrolled patients' post-randomization, either through face-to-face visits or telephone follow-ups.

ELIGIBILITY:
Inclusion Criteria ：

1. . Age 18 to 80 years, any gender.
2. . Clinically confirmed acute spontaneous supratentorial intracerebral hemorrhage (ICH), with diagnostic CT completed within 24 hours of symptom onset (for patients with unknown time of onset or wake-up stroke, the time from the last known well to symptom detection is used as the presumed onset time).
3. . CT-confirmed supratentorial ICH with hematoma volume calculated by ABC/2 method between 25 mL and 60 mL (inclusive).
4. . National Institutes of Health Stroke Scale (NIHSS) score ≥ 6.
5. .Glasgow Coma Scale (GCS) score between 9 and 14 (inclusive).
6. . Pre-stroke modified Rankin Scale (mRS) score ≤ 1.
7. . Good compliance, with written informed consent provided by the patient and/or legal guardian, and ability to adhere to the scheduled follow-up visits.

Exclusion Criteria：

1. . Brainstem or cerebellar hemorrhage; or thalamic hemorrhage with significant midbrain shift accompanied by third nerve palsy or unreactive dilated pupils.
2. . Irreversible brainstem dysfunction (bilateral fixed, dilated pupils and decerebrate posturing).
3. . Secondary ICH caused by: head trauma, arteriovenous malformation (AVM), moyamoya disease, intracranial aneurysm, coagulation disorders (hereditary or acquired hemorrhagic diathesis, hemophilia, coagulation factor deficiency, leukemia, etc.), hemorrhagic transformation of cerebral infarction, or tumor; multiple intracranial hemorrhages, subarachnoid hemorrhage (SAH), primary intraventricular hemorrhage, drug-induced hemorrhagic stroke, subdural hemorrhage, epidural hemorrhage.
4. . Significant abnormalities in the following laboratory parameters:(1)International normalized ratio (INR) > 1.4; any irreversible coagulopathy or known coagulation disorder that cannot be corrected with procoagulants to maintain INR ≤ 1.4. (2) Severe hepatic insufficiency: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 3 times the upper limit of normal (ULN). (3) Severe renal insufficiency: estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m². (4)Hemoglobin < 90 g/L.5）Platelet count < 100 × 10⁹/L.
5. . History of malignancy, autoimmune diseases (including but not limited to systemic lupus erythematosus, systemic vasculitis), hemorrhagic diathesis (including various hereditary and acquired bleeding disorders), malignant arrhythmias, cardiac insufficiency (B-type natriuretic peptide [BNP] ≥ 1000 pg/mL or left ventricular ejection fraction [LVEF] ≤ 40%), acute myocardial infarction, acute or severe infectious diseases (e.g., intracranial infection, severe pneumonia, sepsis), or any other severe concurrent illness that may exacerbate the condition or interfere with efficacy assessment.
6. . Known high risk of thromboembolism, including: presence of a mechanical heart valve prosthesis, history of left heart thrombus, mitral stenosis with atrial fibrillation, acute pericarditis, or subacute bacterial endocarditis. (Note: Atrial fibrillation without mitral stenosis is permitted).
7. . Myocardial infarction within 30 days prior to randomization.
8. .Use of anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, apixaban) within 1 week prior to symptom onset.
9. . History of internal bleeding (e.g., gastrointestinal bleeding, genitourinary bleeding, retroperitoneal bleeding) within 3 months prior to randomization.
10. . Major surgery or vascular puncture (e.g., venesection, arterial puncture) within 3 months prior to randomization.
11. . History of significant head trauma or severe stroke within 3 months prior to randomization.
12. . History of intracerebral hemorrhage within 1 year prior to randomization.
13. . Indications for craniotomy: (1) Progressive impairment of consciousness; (2)Preoperative signs of brain herniation (e.g., foramen magnum herniation, tentorial herniation) posing a life-threatening condition.
14. . Intraventricular hemorrhage (IVH) or ICH with rupture into the ventricle causing intraventricular cast formation and/or hydrocephalus anticipated to require external ventricular drainage (EVD).
15. . Patient or family requests craniotomy or neuroendoscopic surgery for hematoma evacuation.
16. . Pre-randomization decision by patient/family for Do-Not-Resuscitate (DNR) or Do-Not-Intubate (DNI) orders regarding life-sustaining measures.
17. . Known hypersensitivity or intolerance to TNK.
18. . Pregnancy (positive urine pregnancy test) in women of childbearing potential.
19. . Concurrent participation in another investigational drug or device study.
20. . History of drug or alcohol abuse/dependence, severe dementia, or psychiatric disorder prior to randomization, anticipated to result in poor compliance and inability to complete follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 768 (Estimated)
Dates: Start 2025-10-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional Improvement (good functional outcome: mRS 0-3) | 180 days post-randomization
  The primary outcome is the proportion of patients with a favorable functional outcome (mRS score 0-3) at 180 days post-randomization.

SECONDARY OUTCOMES:
Functional Improvement (Ordinal analysis of mRS) | 180 days post-randomization
  Ordinal analysis of mRS scores at 180 days post-randomization
Functional Improvement (uw-mRS) | 180 days post-randomization
  Functional Improvement as determined by utility-weighted modified Rankin Scale (uw-mRS) which is assigned to seven levels: 1.0, 0.91, 0.76, 0.65, 0.33, 0.0, and 0.0 (with higher scores indicating a better outcome, according to patients' assessment)
Functional Improvement (good functional outcome mRS 0-2) | 180 days post-randomization
  Proportion of subjects with mRS score 0-2 at 180 days post-randomization
Functional Improvement (good functional outcome mRS 0-1) | 180 days post-randomization
  Proportion of subjects with mRS score 0-1 at 180 days post-randomization
Functional Improvement (good functional outcome: eGOS 4-8) | 180 days post-randomization
  eGOS score at 180 days post-randomization (favorable: 4-8; unfavorable: 1-3)
Mortality | 180 days post-randomization
  All-cause mortality at 180 days post-randomization
Health-related quality of daily life | 180 days post-randomization
  EQ-5D-5L score at 180 days post-randomization
Early neurological improvement | Day 7 (or at early discharge if earlier)
  Change in NIHSS score from baseline to Day 7 (or at early discharge if earlier)
Residual hematoma volume | Day 7 post-randomization
  Residual hematoma volume on Day 7 post-randomization
Clot removal rate | 7 days post-randomization
  Hematoma clearance rate at 7 days post-randomization
Length of hospital stay and economic | from symptom onset to 180 days post-randomization
  ICU length of stay (from symptom onset to end of follow-up)

OTHER OUTCOMES:
Safety outcome: All-cause mortality within 30 days post-randomization | 30 days post-randomization
  All-cause mortality within 30 days post-randomization is the primary safety outcome
Safety outcome: Symptomatic rebleeding rate within 30 days post-randomization | 30 days post-randomization
  Symptomatic rebleeding rate within 30 days post-randomization
Safety outcome: Bacterial intracranial infection | 30 days post-randomization
  Intracranial infection rate within 30 days post-randomization
Serious Adverse Events | 180 days post-randomization
  Overall incidence of Serious Adverse Events within 180 days post-randomization
Adverse Events | 180 days post-randomization.
  Overall incidence of Adverse Events within 180 days post-randomization.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Suzhou First People's Hospital, Suzhou, Anhui
  - Guizhou Medical University Affiliated Hospital, Guiyang, Guizhou

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP